CLINICAL TRIAL: NCT05626374
Title: A Cluster Randomized, 2x2 Factorial, Superiority Study to Compare the Effectiveness of Adding a Remote Self-reporting Tool for Distress and a Fit-for-purpose Mental Health & Addictions Service to Usual Case Management on Program Completion and Employment Among Unemployed Visible Minorities and Women Enrolled in a Vocational Training Program
Brief Title: Comparing the Effect of Adding a Remote Self-reporting Tool for Distress and Fit-for-purpose Mental Health & Addictions Service to Usual Case Management on Dropout Rates in a Vocational Training Program
Acronym: TeachMeToBuild
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Victoria Hospital, Canada (Other)
Responsible Party: Principal Investigator, Giulio DiDiodato, Chief Research Scientist, Royal Victoria Hospital, Canada
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: R22-013
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Mental Health Issue; Substance Use Disorders; Distress, Emotional
Keywords: mental health issues; substance use disorders; multi-centre trial; cluster randomized; factorial design; vocational training program; vulnerable youth; unemployment
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: 2x2 factorial design, cluster-randomized, multicentre trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Basic case management (Active Comparator): Basic case management with bi-weekly meetings between case manager and trainees that includes check-ins, frequent visits to construction sites and monitoring of feedback forms from mentors. Case managers attempt to connect trainees with external support services as needed.
  Interventions: Behavioral: Basic Case Management
- Basic case management supplemented by self-reporting distress tool (DT) (Experimental): Basic case management plus access to the self-report daily distress tool. The trainees are provided web-based access to the daily distress tool and report their distress levels using a validated visual analog scale (Distress Thermometer), along with reporting their risk of missing work/class or dropping out of the program. The case manager responds to the distress tool by coordinating external support services as needed.
  Interventions: Behavioral: Basic Case Management plus Distress Tool
- Basic case management supplemented by rapid access healthcare services (Experimental): Basic case management supplemented by a fit-for-purpose rapid referral process for trainees with active mental health and/or substance use disorders affecting their program participation.
  Interventions: Behavioral: Basic Case Management plus rapid mental health & addictions healthcare access
- Basic case management supplemented by DT and rapid access healthcare services (Experimental): Basic case management supplemented by both the self-report distress tool and rapid referral process for those trainees at-risk of program absence or drop-out from either mental health or addictions issues.
  Interventions: Behavioral: Basic Case Management plus Distress Tool and rapid mental health & addictions healthcare access

INTERVENTIONS:
Behavioral: Basic Case Management — Usual case management support during 12-week training program
  Arms: Basic case management
Behavioral: Basic Case Management plus Distress Tool — Usual case management support during 12-week training program plus daily self-reports of distress using Distress Thermometer tool
  Arms: Basic case management supplemented by self-reporting distress tool (DT)
Behavioral: Basic Case Management plus rapid mental health & addictions healthcare access — Usual case management support during 12-week training program plus rapid access referral process for healthcare crisis services
  Arms: Basic case management supplemented by rapid access healthcare services
Behavioral: Basic Case Management plus Distress Tool and rapid mental health & addictions healthcare access — Usual case management support during 12-week training program plus daily distress self-reports plus rapid access referral process for healthcare crisis services
  Arms: Basic case management supplemented by DT and rapid access healthcare services

SUMMARY:
Youth unemployment is a chronic problem in most societies. Some young adults are neither in employment, education or training (NEET), and are at high risk of chronic unemployment, social disengagement and poor quality of life. Identifying this high risk population and providing them with career skills training and opportunities is critical for their full participation in society. Vocational training programs provide an opportunity for these NEET youth to develop a skilled trade. Barriers to successful completion of these programs include high prevalence of mental health and substance use disorders among NEET youth. This study will use a daily self-report distress tool to identify vocational program trainees at risk of absence or drop-out due to mental health and/or substance abuse issues. These at-risk trainees will then be referred to a mental health crisis program through a fit-for-purpose referral process to accommodate their training program requirements. It is hypothesized that early identification and referral for mental health and substance abuse issues will reduce both program absence and drop-out rates and result in improved in long-term employment for these NEET youth.

DETAILED DESCRIPTION:
The Trades & Diversity Training Program (TDTP) is a Canadian federal government-funded vocational construction skills training program for visible minority & female youth who are chronically under- and unemployed. The TDTP is a 12-week program that includes both in-classroom education and supervised hands-on experiential learning at participating construction sites. The trainees are supported by a case manager who identifies, plans and co-ordinates support services to minimize program absences and drop-out. The most significant barriers to successful program completion and long-term employment are mental health and substance use disorders. Historically, identification and rapid referral to mental health and addiction services has been difficult due to human resource limitations and limited access to timely healthcare services. This study will randomize cohorts enrolled in each 12-week training program located in 2 sites to the use of a self-report distress tool versus usual case management. The distress tool is a web-based self-reporting tool that is accessed by trainees on a daily basis to report their distress levels, the underlying reasons for this distress and whether this distress will prevent them from attending class or put them at-risk for drop-out. For those individuals whose distress levels threaten their program participation, the case manager is alerted immediately via an email notification. The case manager is then responsible for connecting with the trainees and engaging the rapid referral process for mental health and addictions healthcare services. The control cohorts will receive the usual case management approach of engaging students on an intermittent basis and providing support as needed.

ELIGIBILITY:
Inclusion Criteria:

* must be a visible minority or female
* must be fluent in English or French
* must have an active Ontario Health Insurance Plan number
* must have a valid Canadian Social Insurance Number
* Access to wi-fi network and computing device (phone, tablet, computer)

Exclusion Criteria:

- none

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female based on self-representation of gender identity
Enrollment: 400 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Program attendance | 12 weeks from program enrolment
  Difference in proportion of absence-free program days, where absence-free day is defined as being present in class or work setting by case manager or supervisor. Maximum number of absence-free days is 48 days (12 weeks x 4-day work week). A day is defined as an 8- to 10-hour work day from Monday to Thursday.
Program completion | 12 weeks from program enrolment
  Difference in proportion of drop-outs, where a drop-out is defined as an apprentice who fulfils any of the following criteria:
  1. Has missed more than 50% of class/work days, or
  2. Who has elected to leave the program for reasons other than taking another job or returning to school
Post-program employment | 24 weeks post-program completion
  Difference in proportion of full-time employment, where full-time employment is defined as paid work ≥ 30 (median) hours per week at their main or only job. The reference period that will be used to determine full-time employment is the 4-week period preceding the 24-month post-program completion date.

SECONDARY OUTCOMES:
Access to healthcare services | 12 weeks from program enrolment
  Difference in time to access mental health & addiction services, where time to access is defined as the difference (hours) between the date of referral from the case manager to the date of the mental health & addictions appointment/assessment.
Healthcare utilization | 12 weeks from program enrolment
  Difference in incidence rates of healthcare days, where healthcare days represent the number of days alive and registered for an emergency room, mental health outpatient or addictions outpatient visit, or admitted to an acute care, mental health or detoxification facility. The potential number of healthcare days is the number of days alive during the program (12 weeks x 7 days = 84 days)
Apprentice satisfaction | 12 weeks from program enrolment
  Difference in program satisfaction scores, where program satisfaction scores will be measured using the validated National Centre for Vocational Education Research Student Outcomes Survey Satisfaction scores
Acceptability of self-report distress tool | 12 weeks from program enrolment
  To measure the acceptability of using the Distress Thermometer screening tool by apprentices and the case manager, where acceptability is measured using a validated 2-item questionnaire.
Feasibility of self-report distress tool | 12 weeks from program enrolment
  To measure the feasibility of using the Distress Thermometer screening tool by apprentices and the case manager, where feasibility is measured using a validated 1-item questionnaire.
Compliance of self-report distress tool | 12 weeks from program enrolment
  To measure apprentices' compliance with the Distress Thermometer screening tool, where compliance is defined as the ratio of completed daily screens relative to the total number of program days

CONTACTS AND LOCATIONS:
Overall Officials: Giulio DiDiodato, MD PhD, Principal Investigator — Royal Victoria Regional Health Centre
Locations (1):
- Royal Victoria Regional Health Centre, Barrie, Ontario, Canada

REFERENCES:
- [Derived] Bailey S, Stoner C, Cruise K, DiDiodato G. Protocol for a cluster randomized study to compare the effectiveness of a self-report distress tool and a mental health referral service to usual case management on program completion among vulnerable youth enrolled in a vocational training program. PLoS One. 2024 Aug 1;19(8):e0294806. doi: 10.1371/journal.pone.0294806. eCollection 2024. PMID 39088460